CLINICAL TRIAL: NCT01036230
Title: The Effects of Expectation on Natural and Drug -Induced Rewards
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904397; 04-DA-N397
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-02-25

CONDITIONS: Drug Abuse
Keywords: fMRI; Methylphenidate; Taste; Olfaction; Addiction
MeSH Terms: conditions — Substance-Related Disorders; Anosmia; Behavior, Addictive

STUDY DESIGN:
Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

* Environmental cues frequently induce expectancies in individuals that may strongly influence the actual experience associated with the cue. This has both positive and negative consequences for behavior and decision making. For instance, when an addicted individual experiences cues associated with imminent drug taking, an expectancy of the coming experience is also formed and very likely has an effect on the subsequent experience of the drug.
* Researchers are interested in studying how the brain responds to these kinds of environmental cues and expectancies in order to learn more about addiction and craving in substance-abusing individuals.

Objectives:

* To compare the response to rewards (both drug-related and non-drug-related) in cocaine users and non-using individuals.
* To study the effect of expectation on reward-related (both drug-induced and non-drug-induced) responses and brain activity in cocaine users and non-using individuals.

Eligibility:

-Individuals between 18 and 45 years of age who are regular cocaine users but otherwise healthy, or healthy individuals who are not cocaine users.

Design:

* This study involves two experiments. Participants will be assigned to one or both experiments.
* Participants must not use any drugs for at least 3 days before the visit, may not consume alcohol for 24 hours before the visit, and may not consume caffeinated beverages for 12 hours before the visit. On the day of the visit, participants will provide both urine and breath samples to test for drug/alcohol use.
* Experiment 1: In the MRI scanner, participants will respond to questions and images on a screen, and will receive small amounts of flavored liquid (chocolate or cherry) through a tube in the mouth.
* Experiment 2: In the MRI scanner, participants will respond to questions and images on a screen, and will receive injections of liquid (saline solution or a drug that provides a high similar to cocaine) through an intravenous line. Participants in this experiment will return for follow-up visits and provide urine samples for further study.
* The specific assignment (to Experiment 1 or Experiment 2 or both experiments) will determine the number of study days and follow-up visits required.

DETAILED DESCRIPTION:
Objective: Environmental cues frequently induce expectancies in the course of normal daily life. When an individual smells and sees the coffee before tasting it, an expectancy of the coming experience is formed that influences the actual experience of consuming the coffee. Similarly, when an addicted individual experiences cues associated with imminent drug taking, an expectancy of the coming experience is also formed. This protocol will examine neural responses to cues predictive of a stimulus (neutral or rewarding) and to the subsequent receipt of the predicted stimulus.

Study Population: Study participants will include 18-50 year old, male and non-pregnant female otherwise healthy cocaine dependent individuals and control individuals who have a history of some stimulant use but no history of abuse or dependence on any other drug other than nicotine.

Design: The study will employ fMRI to elucidate the neural underpinnings of reward processing. The rewarding stimuli to be studied will be taste stimuli (small squirt of juice or chocolate) and a drug stimulus (intravenous methylphenidate (IV MPH)). For taste stimuli, cues will vary in sensory modality (visual vs. olfactory) and in novelty (well-known vs. novel). Novel and well-known cue stimuli will be included on each experimental day so the development of expectancy can be studied as the cue-taste pairing is learned and compared to the well-known cue-taste pairing. The MPH/saline injections will receive a written cue.

Outcome Measures: BOLD fMRI signal to reward stimuli will be compared in the various cuing conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALL PARTICIPANTS MUST:

Be between the ages of 18-50.

Be in good health.

Be right-handed.

Like the flavors of cherry Kool-Aid and Hershey's chocolate sauce.

COCAIN DEPENDENT PARTICIPANTS MUST:

Demonstrate that they area cocaine dependent.

Be users of crack cocaine, free base cocaine or intravenous cocaine.

Fe free of dependence on other substances except nicotine.

Be free of abuse of other substances besides marijuana or alcohol.

CONTROL PARTICIPANTS MUST:

Be free of current or past DSM-IVTR substance use disorder except nicotine dependence or past substance abuse diagnosed iwth the single criterion of recurrent substance use in situations in which it is physically hazardous.

EXCLUSION CRITERIA:

Participants will be excluded if they:

Are not suitable to undergo an fMRI experiment due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology or claustrophobia.

Have cardiovascular disease, including but not limited to clinically significant arrhythmia, coronary artery disease and hypertension.

Have coagulopathies, history of or current superficial or deep vein thrombosis, musculoskeletal abnormalities restricting an individual's ability to lie flat for extended periods of time.

Have HIV or syphilis.

Have any neurological illnesses to include, but not limited to, seizure disorders, frequent migraine, multiple sclerosis, movement disorders, or history of head traume, CVA, CNS tumor

Have an abnormality on screening MRI scans that would place the participant at increased risk from blood pressure elevations related to protocol procedures (methylphenidate injections) or would impair the quality of data gathered on the participant.

Have other major medical illnesses likely to interfere with study results or safety of an individual during participation.

Have any current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders, or substance-induced disorders.

Regularly use any prescription, over-the-counter or herbal medication that may alter CNS function, cardiovascular function or neuronal-vascular coupling.

Are actively seeking or engaged in substance abuse treatment.

Are lactating.

Are cognitively impaired or learning disabled.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05-24; Study Completion 2019-02-25

PRIMARY OUTCOMES:
To compare the response to rewards (drug and non-drug related) in cocaine dependent and non- dependent individuals and study the effect of expectation on reward-related (both drug and non-drug induced) subjective responses and neuronal activity.

SECONDARY OUTCOMES:
To compare visual and olfactory cues as they relate to receipt of a non-drug reward. Olfactory cues follow a more direct path into the limbic system and thus, may alter reward system functioning differently than do visual cues.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Jo Salmeron, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Marlatt GA. Cue exposure and relapse prevention in the treatment of addictive behaviors. Addict Behav. 1990;15(4):395-9. doi: 10.1016/0306-4603(90)90048-3. PMID 2248112
- [Background] Childress AR, Hole AV, Ehrman RN, Robbins SJ, McLellan AT, O'Brien CP. Cue reactivity and cue reactivity interventions in drug dependence. NIDA Res Monogr. 1993;137:73-95. PMID 8289929
- [Background] Ito R, Dalley JW, Robbins TW, Everitt BJ. Dopamine release in the dorsal striatum during cocaine-seeking behavior under the control of a drug-associated cue. J Neurosci. 2002 Jul 15;22(14):6247-53. doi: 10.1523/JNEUROSCI.22-14-06247.2002. PMID 12122083